CLINICAL TRIAL: NCT06358469
Title: STRatIfication of Vulvar Squamous Cell Carcinoma by HPV and p53 Status to Guide Excision
Brief Title: STRatIfication of Vulvar SCC by HPV and p53 Status to Guide Excision
Acronym: STRIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Australia New Zealand Gynaecological Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VU2
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Vulvar Squamous Cell Carcinoma
MeSH Terms: interventions — Surgical Procedures, Operative; Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sub-Study A: Active Surveillance (Active Comparator): If the laboratory test results show vulvar cancer is caused by HPV
  Interventions: Other: Active Surveillance
- Sub-Study B: Re-excision (Active Comparator): If the laboratory test results show vulvar cancer is not caused by HPV
  Interventions: Procedure: Surgery
- Sub-Study B: Active Surveillance (Active Comparator): If the laboratory test results show vulvar cancer is not caused by HPV
  Interventions: Other: Active Surveillance

INTERVENTIONS:
Procedure: Surgery — Re-excision of vulvar cancer margin
  Arms: Sub-Study B: Re-excision
Other: Active Surveillance — The investigator will follow the patient to watch for side effects and keep track of patient's health
  Arms: Sub-Study A: Active Surveillance; Sub-Study B: Active Surveillance

SUMMARY:
This study is being done to answer the following question: Are there types of early-stage vulvar cancer that require either less or more treatment than the usual approach?

DETAILED DESCRIPTION:
This study is being done to find out if these approaches are better or worse than the usual approach for early-stage vulvar cancer. The usual approach is defined as care most people get for early-stage vulvar cancer.

The usual approach for patients who are not in a study is treatment with surgery. Tissue that is removed as part of this procedure is analyzed in the pathology laboratory to guide the doctor in deciding whether additional surgery should be recommended.

For patients deciding to take part in this study, the treatment that will be recommended will be based on laboratory testing of the cancer. The laboratory assessments include a test to determine if the cancer is caused by the Human Papilloma Virus (HPV) or not caused by HPV. If the laboratory test results show the vulvar cancer is caused by HPV, the study doctor will recommend the patient participate in sub-study A. In sub-study A, the patient will receive no additional surgery (observation). If the laboratory test results show the vulvar cancer is not caused by HPV, the study doctor will recommend the patient participate in sub-study B. In sub-study B, patients will receive either a second surgery or no additional surgery (observation).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary diagnosis of vulvar squamous cell carcinoma (VSCC)
* Surgically staged FIGO I-II VSCC as per FIGO 2021 guidelines
* Vulvar resection according to standard of care guidelines
* Post-operative margin assessment of tumour clearance, dVIN and p53 status.
* Participants' age must be ≥ 18 years old
* Participant is able (i.e. sufficiently fluent) and willing to complete the quality of life and/or health utility questionnaires in either English or French
* Participant's consent must be appropriately obtained in accordance with applicable local and regulatory requirements

Exclusion Criteria:

* Recurrent vulvar squamous cell carcinoma
* Non-squamous cell carcinoma histotypes
* Participants referred for/receiving/or previously received adjuvant vulvar radiation or chemotherapy
* Primary tumour HPV-I p53 wild-type VSCC
* Surgical margins positive for invasive cancer.
* Participants with a history of other malignancies, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for ≥ 5 years
* Lymph node positive VSCC

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 249 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2031-11-30 (Estimated)

PRIMARY OUTCOMES:
Estimate the 3-year local recurrence rates in patients with HPV-Independent (HPV-I) and HPV-Associated (HPV-A) vulvar squamous cell carcinoma (VSCC) surgically managed based on dVIN/p53 status and tumour margin clearance | 3 years

SECONDARY OUTCOMES:
HPV-I and HPV-A VSCC cohorts: Recurrence-free survival | 3 years
HPV-I and HPV-A VSCC cohorts: Disease-specific survival | 3 years
HPV-I and HPV-A VSCC cohorts: Overall-survival | 3 years
HPV-I and HPV-A VSCC cohorts: Estimate health economic impact of surgical management based on molecular biomarker stratification and margin status assessment utilizing EQ-5D-5L | 3 years
HPV-I and HPV-A VSCC cohorts: Describe patient-reported outcomes utilizing EORTC QLQ-C30 | 3 years
HPV-I and HPV-A VSCC cohorts: Describe patient-reported outcomes utilizing EORTC QLQ-VU34 | 3 years
HPV-I and HPV-A VSCC cohorts: Describe patient-reported outcomes utilizing Fear of Recurrence Scale | 3 years
HPV-I cohort: Estimate recurrence rates of vulvar dVIN and/or p53abn | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Amy Jamieson, Study Chair — University of British Columbia, Vancouver, BC, Canada; Jessica McAlpine, Study Chair — BCCA-Vancouver Cancer Centre, Vancouver, BC Canada
Locations (9):
- Canada (8):
  - BCCA - Vancouver, Vancouver, British Columbia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - CHUM-Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Hotel-Dieu de Quebec, Québec, Quebec
  - CIUSSS de l'Estrie - Centre hospitalier, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
- Auckland City Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No